CLINICAL TRIAL: NCT03277924
Title: Phase I-II Trial of Sunitinib and/or Nivolumab Plus Chemotherapy in Advanced Soft Tissue and Bone Sarcomas
Brief Title: Trial of Sunitinib and/or Nivolumab Plus Chemotherapy in Advanced Soft Tissue and Bone Sarcomas
Acronym: ImmunoSarc
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-52
Record Dates: First submitted 2017-08-03; First posted 2017-09-11 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma
Keywords: Dedifferentiated chondrosarcoma; Extraskeletal myxoid chondrosarcoma; Angiosarcoma; Hemangioendothelioma; Intimal sarcomas; Solitary fibrous tumor; Clear cell sarcoma; Alveolar soft-part sarcoma; Undifferentiated pleomorphic sarcoma; Leiomyosarcoma; Osteosarcoma; Synovial Sarcoma; Epithelioid Hemangioendothelioma; Epithelioid Sarcoma; Ewing's Sarcoma; Chondrosarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Chondrosarcoma, Extraskeletal Myxoid; Hemangiosarcoma; Hemangioendothelioma; Solitary Fibrous Tumors; Sarcoma, Clear Cell; Sarcoma, Alveolar Soft Part; Histiocytoma, Malignant Fibrous; Leiomyosarcoma; Osteosarcoma; Sarcoma, Synovial; Hemangioendothelioma, Epithelioid; Sarcoma, Ewing; Chondrosarcoma | interventions — Sunitinib; Nivolumab; Epirubicin; Ifosfamide; Doxorubicin; Dacarbazine; Cisplatin; Methotrexate

STUDY DESIGN:
Intervention Model Description: Phase I-II, single-arm, non-randomized, open-label, multicenter, international clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sunitinib and/or nivolumab plus chemotherapy in advanced STS and BS (Experimental): Stage 1:
  IP d1-14 sunitinib 37.5mg/d then MP sunitinib 37.5mg/d+nivolumab 3mg/kg ev 2w.
  Stage 2:
  C1-6: IP d1-14 sunitinib 37.5mg/d then MP sunitinib 25mg/d+nivolumab 240mg ev 2w. C7a level 0: Epirubicin 60mg/m2/d, d1,2, ifosfamide 3g/m2/d d1-3 and nivolumab 360mg. 3 or more DLTs level -1 same treatment than in level 0, but nivolumab 240mg. C7b level 0: Doxorubicin 75mg/m2/d, d1, dacarbazine 400mg/m2/d (also on d2) and nivolumab 360mg. 3 or more DLTs level -1 same tratment than in level 0, but nivolumab 240mg. GCSF support is mandatory. 1-year maintenance of nivolumab. C8 level 0: In the IP, CDDP 120mg/m2 (d1-2), doxorubicin 75mg/m2 in (d3-4 and d36-39), nivolumab 240mg (d5), and on d18,39,53 and methotrexate 12g/m2 on d22,29,57,64, surgery and MP with nivolumab on d210, every 2 weeks up to d364. 3 or more DLTs level -1, with nivolumab 360mg on d4,36, surgery and MP with nivolumab on d210, ev 3 weeks up to d364.
  Interventions: Drug: Sunitinib 37.5 MG, Sunitinib 25 MG [Sutent]; Drug: Nivolumab 100 MG/10 ML [Opdivo]; Drug: Epirubicin; Drug: Ifosfamide; Drug: Doxorubicin; Drug: Dacarbazine; Drug: Cisplatin; Drug: Methotrexate

INTERVENTIONS:
Drug: Sunitinib 37.5 MG, Sunitinib 25 MG [Sutent] — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
  Other Names: Sutent
Drug: Nivolumab 100 MG/10 ML [Opdivo] — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
  Other Names: Opdivo
Drug: Epirubicin — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
Drug: Ifosfamide — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
Drug: Doxorubicin — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
Drug: Dacarbazine — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
Drug: Cisplatin — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.
Drug: Methotrexate — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.

SUMMARY:
Phase I-II, single-arm, non-randomized, open-label, multicenter, international clinical trial, with two stages. Stage one has two cohorts (soft tissue sarcoma and bone sarcoma) and stage two has eight cohorts (DDCS, EMC, VS, SFT, CCS, ASPS, UPS, LMS and OS). Nine sites in Spain, 3 sites in Italy and 1 site in the United Kingdom.

Stage 1 (PHASE 1 and PHASE 2)

Objective: To determine the recommended dose of the sunitinib plus nivolumab combination for phase II part. To evaluate the efficacy of the sunitinib plus nivolumab combination as measured by the progression-free survival rate (PFSR) at 6 months in patients with advanced soft tissue and bone sarcomas.

Treatment: Adult patients will receive an initial induction phase (IP) from day 1 to day 14 of sunitinib 37.5 mg/day followed by a maintenance phase (MP) of sunitinib 37.5 mg/day continuously + nivolumab 3 mg/kg intravenous every 2 weeks infused over 1 hour. If three or more DLTs occur from day 15 to 42, for an initial set of 10 patients, sunitinib dose will be lowered to 25 mg/day or treatment schedule will be changed to 2 weeks on and one week off until recovery from toxicities.

Stage 2

C1 to 6

Objective: To evaluate the efficacy of the sunitinib plus nivolumab combination as measured by PFSR at 6 months (CS/DDCS, EMC, VS, SFT, CCS cohorts) and at 12 months (ASPS cohort).

Treatment: Adult patients will receive an initial induction phase (IP) from day 1 to day 14 of sunitinib 37.5 mg/day followed by a maintenance phase (MP) of sunitinib 25mg/day continuously + nivolumab 240mg every 2 weeks. Pediatric patients will receive an initial IP from day 1 to day 14 of (<18 years) sunitinib at 25 mg/day unless the body surface area (BSA) of the patient is >1.7. If BSA is >1.7, then sunitinib 37.5 mg/day will be given followed by a MP of sunitinib 25 mg/day continuously + nivolumab 240 mg every 2 weeks regimen (if weight ≥40 kg) or sunitinib 25 mg/day continuously + nivolumab 3 mg/kg every 2 weeks regimen (if weight <40kg).

C 7

Objective: To determine the MTD of the epirubicin + ifosfamide + nivolumab combination in undifferentiated pleomorphic sarcoma and of the doxorubicin + dacarbazine + nivolumab combination in leiomyosarcoma.

Treatment:Cohort 7a dose level 0: Patients will receive epirubicin dose of 60 mg/m2/d, d1 and d2 IV 20 minutes; followed by ifosfamide 3 g/m2/d d1-3, IV 3h with MESNA protection (40% of total dose of ifosfamide in each administration at 0, 3 and 6 h from ifosfamide initiation). Once finished Ifosfamide infusion of day 3, nivolumab is administered during 30 minutes, at dose of 360 mg IV, Q3W. GCSF support is mandatory. If three or more DLTs occur nivolumab dose will be lowered to dose level -1.

Cohort 7b dose level 0: Patients will receive doxorubicin at dose of 75 mg/m2/d, d1 IV 20 minutes; followed by dacarbazine 400 mg//m2/d IV 60 minutes. Dacarbazine is administered also on day 2 of cycle. Once finished Dacarbazine infusion of day 2, nivolumab is administered for 30 minutes, at dose of 360 mg IV, Q3W. GCSF support is mandatory. If three or more DLTs occur nivolumab dose will be lowered to dose level -1 where patients will receive doxorubicin at dose of 75 mg/m2/d, d1 IV 20 minutes; followed by dacarbazine 400 mg//m2/d IV 60 minutes. Dacarbazine is administered also on day 2 of cycle. Once finished dacarbazine infusion of day 2, nivolumab is administered for 30 minutes, at dose of 240 mg IV, Q3W. GCSF support is mandatory. One-year maintenance of nivolumab is foreseen in the absence of progressive disease.

C 8

Objectives:To determine the MTD of the MAP + nivolumab combination (phase I). Proportion of patients achieving good pathological response (phase II)

Treatment dose level 0: In the IP, patients will receive CDDP 120 mg/m2 in 48h IV infusion (days 1-2) followed by doxorubicin 75 mg/m2 in 48h IV infusion (days 3-4). CDDP and doxorubicin will be given on days 1-4 and 36-39. Nivolumab administration will start on day 4 at flat dose 240 mg (after the end of doxorubicin), being the following doses administered on days 18, 39, and 53 (240 mg). HD methotrexate at 12 g/m2 in 2-h infusion will be administered on days 22, 29, 57, and 64. Surgery will be performed after finishing IP. Adjuvant chemotherapy will be administered after surgery. During the MP patients will receive nivolumab on day 210, every two weeks up to day 364. If three or more DLTs occur, then nivolumab dose level -1 will be activated.

DETAILED DESCRIPTION:
Stage 1

Sample size has been obtained for a one-arm one-stage survival design based on Brookmeyer-Crowley like test. The test statistic for survival probability is assumed to be based on the non-parametric estimate of the survival distribution. For STS 2nd line cohort sample size has been obtained for the primary endpoint progression-free survival rate (PFSR) at 6 months. Estimated accrual time: 24 months. A PFSR of 5% will be considered not promising, whereas a PFSRof 15% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.80, 48 patients are needed in this cohort. For bone sarcoma 2nd line cohort sample size has been obtained under the same assumptions than above, but with a type I error α of 0.10, therefore 38 patients are needed in this cohort.

Stage 2

Cohorts 1-6:

COHORT 1 - Dedifferentiated Chondrosarcoma (DDCS): For DDCS sample size is obtained for the primary endpoint of 6-month progression-free survival rate, estimated accrual 24 months. A 6-m PFSR of 40% will be considered not promising whereas of 70% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 23 patients were estimated in this cohort. With one arm survival design based on survival probability a Brookmeyer-Crowley like test is assumed (Brookmeyer, 1982) [65]. If at least 14 cases over the 23 patients have a 6-m PFSR, then further investigation of the experimental treatment is warranted.

COHORT 2 - Extraskeletal Myxoid Chondrosarcoma (EMC): For EMC sample size is obtained for the primary endpoint of 6-month progression-free survival rate, and estimated accrual 24 months. A 6-m PFSR of 50% will be considered not promising whereas of 80% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 22 patients were estimated in this cohort. With Simon's two-stage Minimax design, at least 13 cases over the 20 first patients (stage 1) should have a 6-m PFSR. Then additional 2 patients would be accrued up to 22 patients. If at least 15 patients had a 6-m PFSR, further investigation of the drug is warranted.

COHORT 3 - Vascular sarcomas (VS) (including angiosarcoma, hemangioendothelioma and intimal sarcomas): For VS sample size is obtained for the primary endpoint of 6-month progression-free survival rate, and estimated accrual 24 months. A 6-m PFSR of 30% will be considered not promising whereas of 60% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 23 patients were estimated in this cohort. With Simon's two-stage Minimax design, at least 8 cases over the 18 first patients (stage 1) should have a 6-m PFSR. Then additional 5 patients would be accrued up to 23 patients. If at least 11 patients had a 6-m PFSR, further investigation of the drug is warranted.

COHORT 4 - Solitary Fibrous Tumor (SFT): For SFT cohort sample size is obtained for the primary endpoint of 6-month progression-free survival rate by Choi criteria, and estimated accrual of 24 months. A 6-m PFSR of 35% will be considered not promising whereas of 65% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 24 patients were estimated in this cohort. With Simon's two-stage Minimax design, at least 6 cases over the 14 first patients (stage 1) should have a 6-m PFSR. Then additional 10 patients would be accrued up to 24 patients. If at least 13 patients had a 6-m PFSR, further investigation of the drug is warranted.

COHORT 5 - Alveolar Soft Part Sarcoma (ASPS): For ASPS cohort sample size is obtained for the primary endpoint of 12-month progression-free survival rate by RECIST criteria, and estimated accrual 24 months. A 12-m PFSR of 40% will be considered not promising whereas of 75% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 18 patients were estimated in this cohort. With Simon's two stage Minimax design, at least 7 cases over the 12 first patients (stage 1) should have a 12-m PFSR. Then additional 6 patients would be accrued up to 18 patients. If at least 11 patients had a 12-m PFSR, further investigation of the drug is warranted.

COHORT 6 - Clear Cell Sarcoma (CCS): For CCS cohort sample size is obtained for the primary endpoint of 6-month progression-free survival rate by RECIST criteria, and estimated accrual 24 months. A 6-m PFSR of 25% will be considered not promising whereas of 55% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 23 patients were estimated in this cohort. With Simon's two-stage Minimax design, at least 4 cases over the 13 first patients (stage 1) should have a 6-m PFSR. Then additional 10 patients would be accrued up to 23 patients. If at least 10 patients had a 6-m PFSR, further investigation of the drug is warranted. An additional 5-7% of patients may be recruited to compensate for potential unevaluable participants.For the variables that follow binomial distributions, like the PFS rate and for the categorical variables, frequencies and percentages will be calculated as well as their confidence interval. If needed, to compare categorical variables both Chi-square test and Fisher's exact test will be performed. Besides, Kaplan-Meier estimations will be used for PFS. Where possible, exploratory analysis will include Cox models to estimate the impact of several factors on PFS.

Cohort 7: This cohort includes a phase 1b study (3+3 design plus expansion cohorts) and therefore no formal sample size has been calculated. Each subcohort (7a: UPS and 7b: LMS) will include between 10 and 20 patients respectively (including the expansions).

Cohort 8: A phase I/II is planned for this cohort. For the phase I part, the safety of the MAP + nivolumab combination will be assessed using a 3+3 design including 6 patients treated at the recommended phase II dose (RP2D). This phase I could include up to 12 patients approximately. Regarding the phase II part, for osteosarcoma with metastasis at presentation and resectable primary tumor, in patients with less than 40 years, sample size is obtained for the primary endpoint of histological response after 2 MAPs of induction. A proportion of 45% of good histological response (≥90% necrosis) will be considered not promising, whereas 68% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.80, 31 patients were estimated in this cohort. With Simon's two-stage Minimax design, at least 7 cases over the 13 first patients (initial part) should have good histological response. Then, additional 18 eligible patients will be accrued up to 31 patients. If at least 19 patients had good histological response, further investigation of the drug is warranted.

ELIGIBILITY:
INCLUSION CRITERIA:

Stage 1

1. Patients must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging tests, etc.) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 18-80 years.
3. Histologic diagnosis of soft tissue sarcoma (undifferentiated pleomorphic sarcoma, synovial sarcoma, alveolar soft part sarcoma, clear cell sarcoma, angiosarcoma, epithelioid hemangioendothelioma, solitary fibrous tumor,epithelioid sarcoma and extraskeletal myxoid chondrosarcoma) or bone sarcoma (osteosarcoma/high grade bone sarcoma, Ewing's sarcoma, chondrosarcoma and dedifferentiated chondrosarcoma) confirmed by central pathology review. Mandatory paraffin embedded tumor blocks must be provided for all subjects without exception for biomarker analysis before treatment (first biopsy) and at end of month 3 or earlier (second biopsy).
4. Metastatic/advanced disease in progression in the last 6 months.
5. Measurable disease according to RECIST 1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. Adequate hepatic, renal, cardiac, and hematologic function.
8. Laboratory tests as follows:

   * Absolute neutrophil count ≥ 1,200/mm³
   * Platelet count ≥ 100,000/mm³
   * Bilirubin ≤ 1.5 mg/dL
   * PT and INR ≤ 1.5
   * AST and ALT ≤ 2.5 times upper limit of normal
   * Creatinine ≤ 1.5 mg/dL
   * Calcium ≤ 12 mg/dL
   * Blood glucose < 150 mg/dL
9. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan.
10. Females of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to enrollment and agree to use birth control measures during study treatment and for 7 months after its completion. Patients must not be pregnant or nursing at study entry. Women/men of reproductive potential must have agreed to use an effective contraceptive method.

INCLUSION CRITERIA 1, 5, 6, 7, 8, 9 AND 10 OF STAGE 1, ARE REPEATED IN ALL COHORTS OF STAGE 2.

Stage 2

Cohort 1-6

2. Age: 12-80 years. 3. Diagnosis of dedifferentiated chondrosarcoma, extraskeletal myxoid chondrosarcoma, vascular sarcomas (including angiosarcoma, hemangioendothelioma and intimal sarcomas), solitary fibrous tumor (excluding dedifferentiated SFT), alveolar soft part sarcoma, and clear cell sarcoma confirmed by central pathology review. 4. Mandatory paraffin embedded tumor blocks must be provided for all subjects without exception for biomarker analysis before treatment. 5. Metastatic/locally advanced unresectable disease in progression in the last 6 months according to RECIST 1.1. Patients with recent diagnosis of metastatic disease can be eligible (if they are not candidates to anthracycline-based treatment).

6. Patients should have previously received at least anthracyclines. Patients in the cohorts of subtypes sensitive to antiangiogenic therapy (SFT, ASPS, CCS, EMC or DDCS) are eligible even if not previously treated. 7. Previous therapy with antiangiogenics is allowed.

Cohort 7

2. Age: 18-80 years. 3. Diagnosis of advanced/metastatic undifferentiated pleomorphic sarcoma (UPS) (cohort 7a) or leiomyosarcoma (LMS) (cohort 7b) confirmed by central pathology review. 4. Mandatory pre-treatment formalin-fixed paraffin embedded (FFPE) tumor tissue must be provided for all subjects without exception for central pathology review and the translational study. Archive tissue can be used for diagnosis confirmation but a recent biopsy (<3 months) is mandatory for translational research. If it is not available or is older than 3 months, the patient must be willing to have a pre-treatment re-biopsy of primary or metastatic tumor (baseline biopsy) within 28 days prior to enrollment. 7. The patient must be naïve of any previous treatment with anthracyclines (not even in adjuvant chemotherapy). 12. Women and men of reproductive potential must have agreed to use an effective contraceptive method during study treatment and for 6 months after the last dose of study drug.

Cohort 8

1. The patient or his/her legal tutors must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow-up. Informed consent must be obtained prior to start of screening process. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging tests, etc.) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 12-40 years.
3. Diagnosis of resectable primary metastatic high-grade osteosarcoma confirmed by central pathology review. Resection of primary tumor +/- metastatic disease has to be feasible and planned.
4. Mandatory pre-treatment formalin-fixed paraffin embedded (FFPE) tumor tissue must be provided for all subjects without exception for central pathology review and the translational study. The patient must be willing to have a pre-treatment re-biopsy of primary or metastatic tumor (baseline biopsy) within 28 days prior to enrollment if diagnosis biopsy does not have enough remaining tissue for translational purposes.

7. The patient must be naïve of any previous treatment. 12. Women and men of reproductive potential must have agreed to use an effective contraceptive method during study treatment and for 6 months after the last dose of study drug.

EXCLUSION CRITERIA:

Stage 1

1. Four or more previous lines of chemotherapy for the advanced disease.
2. Previous anti-programmed death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti PD-L2 or anti CTLA-4 antibody.
3. Prior immune-related adverse event (Grade 3 or higher immune-related pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.).
4. Active, known or suspected autoimmune disease.
5. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI CTCAE version 4.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
7. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
8. Other disease or illness within the past 6 months, including any of the following: • Myocardial infarction Severe or unstable angina • Coronary or peripheral artery bypass graft • Symptomatic congestive heart failure • Cerebrovascular accident or transient ischemic attack • Pulmonary embolism 9. Evidence of a bleeding diathesis. 10. Ongoing cardiac dysrhythmias > Grade 2. 11. Uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg despite optimal medical therapy. 12. Psychiatric illness or social situation that would preclude study compliance. 13. Pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication. 14. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG. 15. Hemorrhage ≥ Grade 3 in the past 4 weeks. 16. History of allergy to study drug components. 17. Previous anticoagulants due to thrombotic events. 18. History of another cancer with the exception of adequately treated basal cell carcinoma or cervical cancer in situ. 19. Presence of brain or central nervous system metastases.

Stage 2

Cohort 1-6

1. Four or more previous lines of chemotherapy.
2. Previous anti-programmed death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti PD-L2 or anti CTLA-4 antibody.
3. Prior immune-related adverse event (Grade 3 or higher immune-related pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.).
4. Active, known or suspected autoimmune disease.
5. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Uncontrolled intercurrent illness (or within 12 months prior to first dose of study drug) including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI-CTCAE] version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
7. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
8. Other disease or illness within the past 12 months, including any of the following:

   * Myocardial infarction
   * Severe or unstable angina
   * Coronary or peripheral artery bypass graft
   * Symptomatic congestive heart failure
   * Cerebrovascular accident or transient ischemic attack
   * Pulmonary embolism
9. Evidence of a bleeding diathesis.
10. Uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg despite optimal medical therapy.
11. Pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication.
12. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
13. Hemorrhage ≥ Grade 3 in the past 4 weeks.
14. History of allergy to study drug components.
15. Anticoagulants due to thrombotic events, with the exception of deep venous thrombosis in limbs, with a stable dose of low-weigh heparine and in the absence of secondary hemorrages.
16. History of another cancer in the previous 5 years with the exception of adequately treated squamous or basal cell carcinoma of the skin or cervical cancer in situ.
17. Presence of brain or central nervous system metastases, unless they are controlled (completely resected or irradiated and/or asympthomatic, no need of steroids).
18. Unwilling to participate in the translational study (not providing mandatory biopsies at baseline).
19. Live vaccine 30 days or fewer prior to enrollment.

Cohort 7

1. Diagnosis of any sarcoma different from undifferentiated pleomorphic sarcoma and leiomyosarcoma.
2. Previous treatment with anthracyclines or any other systemic therapy for advanced sarcoma. The exception is hormone therapy or previous systemic therapy for a previous neoplasm (see exclusion criteria number 13), if this is controlled as long as previous therapy did not include anthracyclines. Adjuvant therapy not containing anthracyclines (eg: gemcitabine-docetaxel) is allowed.
3. Previous anti-programmed death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti PD-L2 or anti CTLA-4 antibody.
4. Prior immune-related adverse event (Grade 3 or higher immune-related pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.).
5. Active, known or suspected autoimmune disease.
6. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI-CTCAE] version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
8. HBV and HCV serologies must be preformed prior to inclusion. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection is not allowed.
9. Pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication.
10. Any of the following diseases/illnesses within the previous 6 months:

    * Myocardial infarction
    * Severe or unstable angina
    * Coronary or peripheral artery bypass graft
    * Symptomatic congestive heart failure
    * Cerebrovascular accident or transient ischemic attack (TIA)
    * Pulmonary embolism
    * Evidence of a bleeding diathesis.
    * Ongoing cardiac dysrhythmias > Grade 2.
11. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
12. History of allergy to study drug components.
13. History of another cancer with the exception of adequately treated basal cell carcinoma or in situ cervical cancer, or with a relapse-free interval longer than 3 years after treatment of the primary cancer with no substantial risk of recurrence.
14. Presence of brain or central nervous system metastases at the time of enrollment, unless they are controlled (completely resected or irradiated and/or asympthomatic, no need of steroids).
15. Patient is unwilling to provide mandatory translational tumor samples or biopsies (if required) cannot be easily traken.

Cohort 8

1. Diagnosis of parosteal, periosteal osteosarcoma or any other bone sarcoma.
2. Previous systemic therapy.
3. Previous anti-programmed death-1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti PD-L2 or anti CTLA-4 antibody.
4. Prior immune-related adverse event (Grade 3 or higher immune-related pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.).
5. Active, known or suspected autoimmune disease.
6. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI-CTCAE] version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
8. HBV and HCV serologies must be performed prior to inclusion. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection is not allowed.
9. Pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication.
10. Any of the following diseases/illnesses within the previous 6 months:

    * Myocardial infarction
    * Severe or unstable angina
    * Coronary or peripheral artery bypass graft
    * Symptomatic congestive heart failure
    * Cerebrovascular accident or transient ischemic attack (TIA)
    * Pulmonary embolism
    * Evidence of a bleeding diathesis
    * Ongoing cardiac dysrhythmias > Grade 2.
11. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
12. History of allergy to study drug components.
13. History of another cancer with the exception of adequately treated basal cell carcinoma or in situ cervical cancer, or with a relapse-free interval longer than 3 years after treatment of the primary cancer with no substantial risk of recurrence.
14. Presence of brain or central nervous system metastases at the time of enrollment, unless they are controlled (completely resected or irradiated and/or asympthomatic, no need of steroids).
15. Patient is unwilling to provide mandatory translational tumor samples or biopsies (if required) cannot be easily taken.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Stage 1 - PHASE 1 | 6 months
  The recommended dose of the sunitinib and nivolumab combination for phase II part will be determined by assessing adverse events according to CTCAE 4.0 and they will be used as a rule for escalating or diminishing dose levels according to the dose-limiting toxicities detailed in the protocol
Stage 1 - PHASE 2 | 6 months
  Progression-free survival rate (PFSR): Efficacy measured by the PFSR at 6 months according to RECIST 1.1. PFSR at 6 months is defined as the percentage of patients who did not experience progression or death due to any cause since enrollment until month 6 after enrollment.
Stage 2 - Cohort 1-6: Progression-free survival rate (PFSR) | 6 months for CS/DDCS, EMC, VS, SFT, and CCS and 12 months for ASPS
  CS/DDCS, EMC, VS, SFT, and CCS cohorts: 6-month progression-free survival rate (PFSR): Efficacy measured by the PFSR at 6 months according to RECIST 1.1. PFSR at 6 months is defined as the percentage of patients who did not experience progression or death due to any cause since enrollmentuntil month 6 after enrollment.
  ASPS cohort: 12-month progression-free survival rate (PFSR): Efficacy measured by the PFSR at 12 months according to RECIST 1.1. PFSR at 12 months is defined as the percentage of patients who did not experience progression or death due to any cause since the date of enrollment until month 12 after enrollment.
Stage 2 - Cohort 7: Maximum tolerated dose (MTD) | 1 year
  The maximum tolerated dose (MTD) of the epirubicin + ifosfamide + nivolumab combination will be determined by assessing adverse events according to CTCAE 5.0 and they will be used for adjusting dose levels according to the dose-limiting toxicities detailed in the protocol.
Stage 2 - Cohort 8: Maximum tolerated dose (MTD) | 1 year
  The maximum tolerated dose (MTD) of the MAP + nivolumab combination will be determined by assessing adverse events according to CTCAE 5.0 and they will be used for adjusting dose levels according to the dose-limiting toxicities detailed in the protocol.

SECONDARY OUTCOMES:
Stage 1 and Stage 2 - Overall survival (OS) | 2 years
  OS is defined as the time between the date of enrollment and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Stage 1 and Stage 2 - Objective response rate (ORR) | 2 months
  ORR is defined as the number of subjects with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) divided by the number of response evaluable subjects (according to RECIST 1.1 criteria).
Stage 2 - Cohort 1-6 Correlation between efficacy and potential predictive biomarkers | 2 years
  Assessed by finding relationships between clinical efficacy results and translational data.
Stage 1 and Stage 2 - Safety profile: Adverse events | 3 years
  Safety profile of the experimental treatment, through assessment of adverse event type, incidence, severity, time of appearance, related causes, as well as physical explorations and laboratory tests. Toxicity will be graded and tabulated by using CTCAE 5.0.
Stage 1 (PHASE 2) and Stage 2 - Cohort 1-6 Clinical outcome | At 36 months
  Clinical outcomes of post protocol treatments assessed by observation of such treatments in follow-up stage.
Stage 2 - Cohort 1-6 Prognostic and response correlation | 1 month
  Prognostic and response correlation with neutrophils/platelets; lymphocytes/platelets; andred blood cell distribution width (RDW), by assessing hematology tests at baseline, after 2 weeks (before nivolumab), after 1 month, at progression, and at response.
Stage 1 (PHASE 1) and Stage 2 - Cohort 1-6 6-month progression-free survival rate (PFSR) | 6 months
  Efficacy measured by the PFSR at 6 months according to RECIST 1.1. PFSR at 6 months is defined as the percentage of patients who did not experience progression or death due to any cause since the date of enrollment until month 6 after enrollment.
Stage 2 - Cohort 7 Median progression-free survival (mPFS) | 6 months
  PFS is defined as the time between the date of enrollment and the date of progression or death due to any cause.
Stage 2 - Cohort 7 Median overall survival (mOS) | 2 years
  OS is defined as the time between the date of enrollment and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Stage 2 - Cohort 8 Pathological response | At month 3
  Measured by percentage of necrosis in surgical specimen.
Stage 1 (PHASE 2) | 3 years
  Efficacy measured through tumor response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow up until tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín Broto, Study Director — Hospital Universitario Fundación Jiménez Díaz; Andrés Redondo, Principal Investigator — Hospital Universitario La Paz; Claudia Valverde, Principal Investigator — Hospital Universitari Vall d'Hebrón; Antonio López Pousa, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Roberto Diaz de Beveridge, Principal Investigator — Hospital Universitario La Fe; Javier Martínez Trufero, Principal Investigator — Hospital Miguel Servet; Irene Carrasco, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Enrique González, Principal Investigator — Hospital Universitario 12 de Octubre; Josefina Cruz, Principal Investigator — Hospital Universitario de Canarias; Silvia Stacchiotti, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Giovanni Grignani, Principal Investigator — Candiolo Cancer Institute - FPO, IRCCS; Emanuela Palmerini, Principal Investigator — Istituto Ortopedico Rizzoli; Sandra Strauss, Principal Investigator — University College London Hospitals; Cristina Mata, Principal Investigator — Hospital General Universitario Gregorio Marañón; Antonio Casado, Principal Investigator — Hospital Clínico Universitario San Carlos; Alejandro Pérez Fidalgo, Principal Investigator — Hospital Clínico Universitario de Valencia; Luis De Sande, Principal Investigator — Hospital Universitario de León; Alba Rubio, Principal Investigator — Hospital Infantil Universitario Niño Jesús; Jerónimo Martínez, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (13):
- Italy (3):
  - Istituto Ortopedico Rizzoli, Bologna
  - Candiolo Cancer Institute - FPO, IRCCS, Candiolo
  - Istituto Nazionale dei Tumori, Milan
- Spain (9):
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Martin-Broto J, Diaz-Beveridge R, Moura D, Ramos R, Martinez-Trufero J, Carrasco I, Sebio A, Gonzalez-Billalabeitia E, Gutierrez A, Fernandez-Jara J, Hernandez-Vargas L, Cruz J, Valverde C, Hindi N. Phase Ib Study for the Combination of Doxorubicin, Dacarbazine, and Nivolumab as the Upfront Treatment in Patients With Advanced Leiomyosarcoma: A Study by the Spanish Sarcoma Group (GEIS). J Clin Oncol. 2025 Jan 20;43(3):297-307. doi: 10.1200/JCO.24.00358. Epub 2024 Oct 2. PMID 39356980
- [Derived] Martin-Broto J, Hindi N, Grignani G, Martinez-Trufero J, Redondo A, Valverde C, Stacchiotti S, Lopez-Pousa A, D'Ambrosio L, Gutierrez A, Perez-Vega H, Encinas-Tobajas V, de Alava E, Collini P, Pena-Chilet M, Dopazo J, Carrasco-Garcia I, Lopez-Alvarez M, Moura DS, Lopez-Martin JA. Nivolumab and sunitinib combination in advanced soft tissue sarcomas: a multicenter, single-arm, phase Ib/II trial. J Immunother Cancer. 2020 Nov;8(2):e001561. doi: 10.1136/jitc-2020-001561. PMID 33203665
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903